CLINICAL TRIAL: NCT02358655
Title: Canadian Community Utilization of Stroke Prevention Study - Emergency Department
Acronym: C-CUSP ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C-CUSP ED
Record Dates: First submitted 2015-01-06; First posted 2015-02-09 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Oral anticoagulant; Knowledge translation; Emergency department
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1: Retrospective Chart Review (Other): Retrospective chart review of all patients who presented to the emergency department (ED) with ECG-documented AF during 1 year prior to study commencement. The main purpose of Phase 1 is to determine if oral anticoagulants were prescribed for eligible AF patients at ED discharge.
  Interventions: Other: Retrospective review of OAC prescription
- Phase 2: Low-Intensity Intervention (Other): Low-intensity intervention will be applied in the ED during 6 months, involving physician education, distribution of an AF patient education package, short-term oral anticoagulant prescription, and a follow-up letter to the patient's family physician.
  Interventions: Other: Prescription of OAC in ED
- Phase 3: High-Intensity Intervention (Other): Phase 3 incorporates the Phase 2 intervention, and adds immediate follow-up (within 48-72 hours) in a community AF clinic run by a nurse/pharmacist who is supervised by a specialist in AF.
  Interventions: Other: Prescription of OAC in ED; Other: Community AF clinic

INTERVENTIONS:
Other: Retrospective review of OAC prescription
  Arms: Phase 1: Retrospective Chart Review
Other: Prescription of OAC in ED
  Arms: Phase 2: Low-Intensity Intervention; Phase 3: High-Intensity Intervention
Other: Community AF clinic
  Arms: Phase 3: High-Intensity Intervention

SUMMARY:
Atrial fibrillation (AF) is a common heart condition, and increases the risk of stroke by six times. There are several medications (blood thinners) that can prevent strokes in AF patients. Many AF patients present to the emergency department, but about half of AF patients leave without prescription of a blood thinner. The study aims to evaluate if adding options like giving a patient education kit, encouraging emergency room physicians to prescribe a blood thinner and providing a specialized AF clinic to patients will increase the number patients receiving blood thinners to prevent strokes.

DETAILED DESCRIPTION:
This is a knowledge translation study will occur in three consecutive phases: Phase 1 is a retrospective chart review of all patients who presented to the emergency department (ED) with ECG documented AF during 1 year prior to study commencement. The main purpose of Phase 1 is to determine if oral anticoagulants (OACs) were prescribed for eligible AF patients at ED discharge. In Phase 2 a low-intensity intervention will be applied in the ED during 6 months, involving physician education, distribution of an AF patient education package, short-term OAC prescription, and a follow-up letter to the patient's family physician. After a one month transition phase, a high intensity intervention will be applied during 6 months in Phase 3. Phase 3 incorporates the Phase 2 intervention, and adds immediate follow-up (within 48-72 hours) in a community AF clinic run by a nurse/pharmacist who is supervised by a specialist in AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the emergency department with electrocardiographically documented atrial fibrillation on a 12 lead ECG

Exclusion Criteria:

* Prosthetic or mechanical mitral or aortic valve
* Known rheumatic heart disease
* Unable to provide informed consent
* Will be admitted to hospital
* Life expectancy of < 6 months
* Metastatic malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
New OAC Prescription (Phase 1 and 3 comparison) | Up to 72 hrs

SECONDARY OUTCOMES:
New OAC Prescription (Phase 1 and 2 comparison) | Up to 72 hrs
New OAC Prescription (Phase 2 and 3 comparison) | Up to 72 hrs
OAC use in eligible patients at 30 days (Phase 2 and 3 comparison) | 30 days
OAC use in eligible patients at 6 months (Phase 2 and 3 comparison) | 6 months
Uptake of study interventions | 6 months
  This outcome measure is meant to determine feasibility for a larger community cluster RCT. This will be measured by the uptake of the interventions described in this study, including: patient use of the AF educational kit, patient use of AF clinic, attendance at educational presentations for patients, family doctors and emergency physicians, patient use of automated text or email reminders for OACs.

OTHER OUTCOMES:
Safety related to OAC, as measured by rates of adverse events related to OAC including major bleeding and minor bleeding | 6 months
  Rates of adverse events related to OAC including major bleeding and minor bleeding will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD, Principal Investigator — Dalhousie University
Locations (5):
- Canada (5):
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick
  - Dartmouth General Hospital, Dartmouth, Nova Scotia
  - Cobequid Community Health Centre, Halifax, Nova Scotia
  - Halifax Infirmary, Halifax, Nova Scotia

REFERENCES:
- [Derived] Parkash R, Magee K, McMullen M, Clory M, D'Astous M, Robichaud M, Andolfatto G, Read B, Wang J, Thabane L, Atzema C, Dorian P, Kaczorowski J, Banner D, Nieuwlaat R, Ivers N, Huynh T, Curran J, Graham I, Connolly S, Healey J. The Canadian Community Utilization of Stroke Prevention Study in Atrial Fibrillation in the Emergency Department (C-CUSP ED). Ann Emerg Med. 2019 Apr;73(4):382-392. doi: 10.1016/j.annemergmed.2018.09.001. Epub 2018 Oct 26. PMID 30502307